CLINICAL TRIAL: NCT06657235
Title: Improved Risk Factor Control Through a Transitional Care Program for Stroke Survivors
Brief Title: Transitional Care Program to Improve Risk Factors in Stroke Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Syntrillo, Inc (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024002
Record Dates: First submitted 2024-10-15; First posted 2024-10-24 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Stroke, Ischemic
Keywords: transitional care program; secondary stroke prevention; stroke care
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Enrollment (Experimental): Participants enrolled around the time of discharge from the hospital immediately following an ischemic stroke.
  Interventions: Other: Transitional Care Program
- Late Enrollment (Experimental): Participants enrolled mainly between 3-5 months after their discharge from the hospital following an ischemic stroke.
  Interventions: Other: Transitional Care Program

INTERVENTIONS:
Other: Transitional Care Program — Participants will receive personalized risk-factor management stroke care from a multidisciplinary team trained by our neurologists to understand the needs of stroke survivors and the nuances of stroke care. Risk factor data from in-home devices, health records, and self-reports will be collected along with functional status and behavioral data obtained through validated questionnaires and an occupational therapy evaluation. Syntrillo's neurology provider will review this data, assess the participant through a telemedicine encounter, and create a comprehensive secondary prevention plan to supplement the participant's care plan at discharge. Data generated through these clinical encounters will be de-identified and used for subsequent development of Syntrillo's stroke management technology.

SUMMARY:
The goal of this clinical trial is to evaluate whether our transitional care program helps stroke survivors better manage their risk factors for stroke to lower the risk of a repeat stroke. The main question it aims to answer is:

- Does the program help participants meet the targets set by the American Heart Association clinical guidelines for control of risk factors associated with stroke?

Researchers will compare participants enrolled right after being discharged from the hospital to participants enrolled around 3-5 months after being discharged to examine whether timing differences in enrollment affect the efficacy of the program.

Participants will:

* Keep track of their medications, their exercise, and their health information using smart devices provided by the study
* Answer questions about their health and lifestyle
* Meet with our team of healthcare providers

ELIGIBILITY:
Inclusion Criteria:

All Cohorts:

* Age 30 or above
* Evidence of ischemic stroke documented on CT or MRI
* Modified Rankin score of 3 or less

Early Enrollment:

* Admission for ischemic stroke at a participating site
* Enrolled during their admission for ischemic stroke or within 24 hours of discharge

Late Enrollment:

* Stroke survivors previously admitted at the participating sites' inpatient stroke unit
* Enrollment date between 1 and 6 months after discharge for inpatient admission for ischemic stroke

Exclusion Criteria:

* Participants determined to have hemorrhagic or periprocedural stroke based on hospital EMR review will be excluded.
* Participants determined to have an ischemic stroke due to dissection based on hospital EMR review will be excluded.
* Participants who lack capacity determined by the care team during their hospitalization (for the early enrollment group) or their most recent clinical encounter (for the late enrollment group) will be excluded.
* Participants with a diagnosis of dementia will be excluded.
* Participants with acute subdural hemorrhage will be excluded.
* Participants with hemorrhagic stroke due to vascular abnormality (aneurysm or AVM) or trauma will be excluded.
* Participants who cannot perform the following will be excluded:

  1. offer a consistent choice about participating in the study
  2. demonstrate that they can comprehend and recall major features of the study including: participation is voluntary, the major procedures, the primary risk, and the primary benefit.
* Participants who are discharged to Long-term Acute Care Hospitals will be excluded.
* Participants who are unable to read or communicate fluently in English will be excluded.
* Participants who do not have reliable internet access to complete telemedicine visits per self-report will be excluded.
* Participants already enrolled in another clinical study which could impact the frequency of monitoring or care that participant receives.
* Participants who do not reside in Virginia, West Virginia, Tennessee, Oklahoma, Illinois, or Michigan will be excluded.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Increased compliance with therapeutic standards of care according to the American Heart Association (AHA) guidelines for secondary stroke prevention in early vs late group | From enrollment to the end of the 6 month monitoring period
  We will measure percent compliance with AHA therapeutic standards in the early enrollment group compared to the anticipated baseline percent compliance in the late enrollment group at equivalent time points post-discharge. Percent compliance is a composite endpoint. Participants will be considered "compliant" to secondary stroke prevention guidelines if all other conditions below (2-5) are met. Participants will be considered "non-compliant" to secondary stroke prevention guidelines if one or more conditions are not met.
90% of systolic blood pressure (SBP) readings < 130 mmHg AND 90% of diastolic blood pressure (DBP) readings < 80 mmHg in a one week period | From enrollment to the end of the 6 month monitoring period
  Blood pressure will be measured using Tenovi's FDA-cleared, portable home blood pressure monitoring device. Both systolic and diastolic measurements must be below the threshold in order for the condition to be met.
Moderate intensity activity > 150 minutes per week on average | From enrollment to the end of the 6 month monitoring period
  Physical activity will be assessed through a combination of self-reported and biometric data. We will administer a physical activity questionnaire and correlate self-reported activity with biometric data obtained from the smartwatch to estimate physical activity and assess confidence level in the data.
Correct prescription of antiplatelet, anticoagulant, and statin medications per guidelines when no contraindications are present | From enrollment to the end of the 6 month monitoring period
  We will verify correct prescriptions and dosing through EHR records, pharmacy records, and/or patient self-report as applicable. Correct prescription and dosing will be determined through expert opinion following AHA therapeutic standards.
Adherence of antiplatelet, anticoagulant, and statin medications > 90% | From enrollment to the end of the 6 month monitoring period
  Adherence is determined by percent of missed doses per week. Medication adherence will be monitored through a combination of self-report, device data, and pharmacy records, as applicable. We will administer the 5-Item Medication Adherence Report Scale (MARS-5) and correlate self-reported data with device data from Tenovi's smart pillbox and pharmacy records to estimate percent adherence and assess confidence level in the data.

SECONDARY OUTCOMES:
Average change in compliance percentage at 1, 2, and 3 months following initiation of our transitional care program | From enrollment to the end of the 6 month monitoring period
  Compliance percent is measured based on the data collected from the four primary outcome measures as described in the primary outcomes.
Frequency of recurrent stroke in the early enrollment cohort compared to the late enrollment cohort at equivalent time points post-discharge | From enrollment to the end of the 6 month monitoring period
  Highest risk for recurrent stroke is in the initial 6 months following the first stroke. Frequency of recurrent stroke will be measured by aggregating the number of patients readmitted to the hospital within 6 months following enrollment based on EHR records and/or patient self-report.
Frequency of readmission in the in the early enrollment cohort compared to the late enrollment cohort at equivalent time points post-discharge | From enrollment to the end of the 6 month monitoring period
  Highest risk for recurrent stroke is in the initial 6 months following the first stroke. Frequency of recurrent stroke will be measured by aggregating the number of patients readmitted to the hospital within 6 months following enrollment based on EHR records and/or patient self-report.

CONTACTS AND LOCATIONS:
Locations (1):
- Valley Health System, Winchester, Virginia, United States

IPD SHARING:
Plan to Share IPD: No